CLINICAL TRIAL: NCT02686125
Title: Prospective Study of Deep Brain Stimulation With the VERCISE™ System for Treatment of Dystonia
Brief Title: Vercise™ DBS Dystonia Prospective Study
Status: Recruiting | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: A4012
Record Dates: First submitted 2016-02-10; First posted 2016-02-19 (Estimated); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Dystonia
MeSH Terms: conditions — Dystonia | interventions — Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Deep Brain Stimulation (DBS) — Subjects receiving Deep Brain Stimulation (DBS) for the treatment of their dystonia symptoms will be offered participation in this registry.
  Other Names: Vercise DBS System Boston Scientific

SUMMARY:
To compile characteristics of real-world outcomes of Boston Scientific Corporation's commercially approved VerciseTM Deep Brain Stimulation (DBS) Systems for the treatment of dystonia.

DETAILED DESCRIPTION:
To compile characteristics of real-world outcomes of Boston Scientific Corporation's commercially approved VerciseTM Deep Brain Stimulation (DBS) Systems for the treatment of dystonia.

Subjects' improvement in disease symptoms and overall Quality of life will be assessed.

ELIGIBILITY:
Inclusion Criteria (IC):

* IC1. Meets criteria established in the locally applicable Vercise System Directions for Use (DFU) for dystonia.
* IC2. At least 7 years old. Parent or guardian consent is required in patients who are younger than 18 years at the time of consent.

Exclusion Criteria (EC):

* EC1. Meets any contraindication in the Vercise System locally applicable Directions for Use.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with intractable primary and secondary dystonia, for persons 7 years of age and older.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-03-07 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with reduction in dystonia symptoms as assessed by BFMDRS score | up to 3 years
Proportion of cervical dystonia subjects with reduction in symptoms as assessed by TWSTRS score | up to 3 years

OTHER OUTCOMES:
Change in SF-36v2 score after DBS (SF-10v2 in patients under the age of 18 years at the time of consent) | upto 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Bloom Lyons, Study Director — Boston Scientific Neuromodulation Corporation
Locations (36):
- Belgium (2):
  - AZ Sint-Lucas, Ghent
  - UZ Gasthuisberg, Leuven
- Queen Elizabeth II Health Sciences Center, Halifax, Canada
- Germany (12):
  - University Berlin, Charite Virchow Standort, Wedding, Berlin
  - Uniklinik Köln, Cologne
  - Universitaetsklinikum Dusseldorf, Düsseldorf
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Universitaetsklinik Eppendorf, Hamburg
  - St. Barbara-Klinik Hamm-Heessen, Hamm
  - Medizinische Hochschule Hannover MHH, Hanover
  - Universitatsklinikum Campus Kiel, Kiel
  - Johannes Gutenberg Universitaet Mainz, Mainz
  - Universitaetsklinikum Giessen und Marburg GmbH, Marburg
  - Evangelisches Krankenhaus Oldenburg, Oldenburg
  - Universitaetsklinikum Wuerzburg, Würzburg
- Medical School of University PECS, Pécs, Hungary
- Hadassah Hebrew University Medical Center, Jerusalem, Israel
- Italy (4):
  - Azienda Ospedaliero-Universitaria di Ferrara, Ferrara
  - Ospedale Dell Angelo, Mestre
  - Policlinico Universitario Agostino Gemelli, Rome
  - Osp. S. Maria Della Misericordia, Udine
- Haga Ziekenhuis locatie Leyweg, The Hague, Netherlands
- Poland (4):
  - 10 Military Clinical Hospital Bydgoszcz, Bydgoszcz
  - Wojewodzki Szpital Dzieciecy Jozefa Brudzinskiego (Childrens Hospital Bydgoszcz), Bydgoszcz
  - Podmiot Leczniczy Copernicus Sp. z o.o., Gdansk
  - Centrum Onkologii - Instytut im. Marii Sklodowskiej-Curie, Warsaw
- National Scientific Center of Neurosurgery N.N. Burdenko, Moscow, Russia
- St. Mary's Hospital Incheon, Incheon, South Korea
- Spain (4):
  - Hospital Clinic de Barcelona, Barcelona
  - University Hospital Virgen Arrixaca, El Palmar
  - Centro Especial Ramon y Cajal, Madrid
  - Hospital General De Asturias, Oviedo
- United Kingdom (4):
  - Southmead Hospital Bristol, Bristol
  - Queen Elizabeth University Hospital, Glasgow
  - Charing Cross Hospital, London
  - Royal Victoria Infirmary, Newcastle upon Tyne